CLINICAL TRIAL: NCT05902338
Title: Motor Skills in Children With Attention Deficit and Hyperactivity Disorder
Brief Title: Effects of Music on Motor Skills of Children With Attention Deficit and Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Zehra Güçhan, PT Assoc Prof, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETK2023
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with music (Experimental): "L400 Over Ear Music Headset Glowing Cat Ear Headphones 7" branded headphones will be used for music intervention.
  Interventions: Other: Music
- Group without music (No Intervention): Music will not be used while performing motor skills.

INTERVENTIONS:
Other: Music — "L400 Over Ear Music Headset Glowing Cat Ear Headphones 7" branded headphones will be used for musical measurements (70-80 bpm music).
  Arms: Group with music

SUMMARY:
Physiotherapists have positive effects on motor skills, executive functions and symptoms of children with attention deficit and hyperactivity disorder. However, progression takes time due to the symptoms of the disease. Physiotherapists need strategies to manage the symptoms of ADHD. Music can be used as a strategy because music is known to reduce the symptoms of children in this group. There is no study in the literature on how motor skills will be affected with musical accompaniment. The aim of this study is to compare motor skills performed with and without music in children with ADHD. When we evaluate motor skills like in a treatment session, the usability of music as an environmental factor will be investigated according to the positive, negative or ineffective results of the music effect.

DETAILED DESCRIPTION:
The American Psychiatric Association defines attention deficit and hyperactivity disorder (ADHD) as one of the most common mental disorders affecting children and adults. The etiology of ADHD is not fully known. Attention deficit, hyperactivity and/or impulsivity are seen as the main symptoms of ADHD. ADHD is grouped into three subtypes according to these symptoms. These three subtypes consist of attention-deficit-dominant type, hyperactivity-dominant type, and combined type with both hyperactivity and inattention symptoms. Researchers reported that 45-70% of children with ADHD have problems in fine and gross motor skills. It is known that problems in motor skills are associated with main symptoms. Balance, gait and postural control are affected in terms of gross motor skills. It has been observed that they perform more slowly in activities that require fine motor skills such as cutting, doing crafts or drawing, and in consecutive finger movements. In addition, handwriting disorders such as dysgraphia are seen in 70% of children with ADHD. During the dual tasks, the sources of attention are divided. Due to this division, the secondary task affects postural performance.

Music is one of the therapy options in some conditions and known as music therapy. It is used in many diseases and conditions such as dementia-alzamer, autism, cerebral palsy, cancer, prematurity, depression and ADHD. Now that music is known to reduce the symptoms of children with ADHD, physical therapists may use music as a strategy. Thus, the purpose of this study is to compare motor skills of children with ADHD with and without music conditions.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with ADHD combined type by a child psychiatrist
* Having adequate cognitive skills to understand the commands of the physiotherapist

Exclusion Criteria:

* Having hearing and/or vision problems
* Having any neurological and/or orthopedic problems that would prevent him from performing the tests
* Having a psychiatric disorder other than ADHD

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Static balance | change from baseline to after 30-minute from the first measurement
  Stork static balance test will be used. Children will be asked to stand comfortably on both feet with their hands on their hips. They will then be asked to raise their non-dominant legs. This test will be repeated 3 times. The test will be measured in time (seconds) with a stopwatch and the best result from three attempts will be recorded.

SECONDARY OUTCOMES:
Dynamic balance | change from baseline to after 30-minute from the first measurement
  Timed up and go (TUG) test will be used. The TUG test is administered using 2 standard chairs and children are asked to walk in a self preferred speed. Time is recorded in seconds.
Nine hole peg test | change from baseline to after 30-minute from the first measurement
  The test consists of a square board with 9 holes. First, the child will be asked to insert the nails into the holes as quickly as possible using the dominant hand, and to quickly remove all the nails from the holes as soon as they are all inserted. Insertion, removal and total time of nails will be recorded in seconds via stopwatch.
Blocking with jenga game | change from baseline to after 30-minute from the first measurement
  Jenga game involves attention and hand eye coordination. The children will be asked to make a standard shape made using six of the game's blocks and the completion time will be recorded in seconds.
Puzzle game | change from baseline to after 30-minute from the first measurement
  A standard wood puzzle will be used to test fine motor skills. The time to complete the puzzle will be recoded in seconds with a stopwatch.
Bruininks-Oseretsky Test of Motor Proficiency-Brief Form (BOTMP-BF) | change from baseline to after 30-minute from the first measurement
  It consists of composite scores of fine motor control, manual coordination, body coordination, strength and agility motor domain. Scoring is done for each subheading. The maximum score that can be obtained from the entire test is 88.
Dual task skill | change from baseline to after 30-minute from the first measurement
  Dual task is based on distraction while doing two tasks at the same time. Performance decreases in dual tasks due to sharing of attention. For the dual task, the child will carry a water filled bottle (500 ml) in his dominant hand while performing the 10-meter walking test. The dual duty will be calculated with the dual duty cost formula. This formula is as follows;
  Dual Task Cost = ((Dual Task Performance - Single Task Performance) X 100/Single Task Performance) The number from calculation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ZEHRA G TOPCU, Principal Investigator — PT. Assoc. Prof.
Locations (1):
- Private clinics, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No